CLINICAL TRIAL: NCT03246698
Title: The Effect of Isolytic and Static Stretching Training in Individuals Having Subacromial Impingement Syndrome With Glenohumeral Internal Rotation Deficit
Brief Title: The Effect of Isolytic and Static Stretching Training in Individuals With Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Halime Ezgi TÜRKSAN, Research Assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3413-GOA
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Shoulder pain; Physical therapy; Rehabilitation; Ultrasonography
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: There are 3 groups. First group will receive isolytic stretching in modified cross body stretching position and standard physiotherapy program. Second group will receive static stretching in modified cross body stretching position and standard physiotherapy program. Control group will receive only standard physiotherapy program. In standard physiotherapy program, there are TENS, hotpack, posture and strengthening training program. Treatment program will last four weeks.
Who Masked: Participant
Masking Description: All of participants must have subacromial impingement syndrome with glenohumeral internal rotation deficit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Isolytic stretching group (Experimental): The participants in this group will receive isolytic stretching in modified cross body position. Additionally they will receive standard physiotherapy.
  Interventions: Other: Isolytic Stretching group
- Static stretching group (Experimental): The participants in this group will receive static stretching in modified cross body position.
  Additionally they will receive standard physiotherapy.
  Interventions: Other: Static Stretching group
- Control group (Active Comparator): The participants in this group will receive only standard physiotherapy.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Isolytic Stretching group — In modified cross body position, isolytic stretching exercises will perform five times each for 15 seconds. After each stretching patient will rest for 5 seconds. When the patient contracts the agonist muscle group with 20% muscle force, the agonist muscle group is stretched at the same time for 2-4 seconds. Isolytic stretching exercises will perform four times a week for four weeks. It's obligatory to receive at least 15 sessions in total. They will also receive standard physiotherapy program four times a week for four week, 15 sessions in total.
  Other Names: Standard physiotherapy
  Arms: Isolytic stretching group
Other: Static Stretching group — In modified cross body position, active-assistive static stretching exercises will be performed 5 times each for 15 seconds. This stretching exercise is performed 5 times with 5 seconds intervals. Static stretching exercises will perform four times a week for four weeks. It's obligatory to receive at least 15 sessions in total. They will also receive standard physiotherapy program four times a week for four week, 15 sessions in total.
  Other Names: Standard physiotherapy
  Arms: Static stretching group
Other: Control group — They will receive only standard physiotherapy program, four times a week for four weeks, 15 sessions in total.
  Other Names: Standard physiotherapy
  Arms: Control group

SUMMARY:
The purpose of this study is to investigate and compare the effect of isolytic and static stretching training in individuals having subacromial impingement syndrome with glenohumeral internal rotation deficit. Isolytic group will receive isolytic stretching in modified cross body stretching position and standard physiotherapy program. Static group will receive static stretching in modified cross body stretching position and standard physiotherapy program. Control group will receive only standard physiotherapy program.

DETAILED DESCRIPTION:
The effectiveness of static stretching on various parameters such as range of motion or pain is studied and proved in literature. Static stretching in cross body position was also found helpful for improving shoulder range of motion with some disadvantages. In modified cross body position, the patient is positioned in a more advantageous way for him/her. Usually this stretching is done as active-assistive static stretching with the physiotherapist. Proof is still needed for the effectiveness of active-assistive static stretching in modified cross body position. Furthermore, there is no research about the effect of isolytic stretching which is relatively new technique compare to static stretches in subacromial impingement syndrome. In isolytic stretching, when the patient contracts the agonist muscle group with 20% muscle force active-assistive streching in agonist muscle group by the physiotherapist at the same time is done for 2-4 seconds. A fast isolytic stretching is applied in order to break the fibrous tissue. Our purpose is to investigate and compare the effect of isolytic and static stretching training in individuals having subacromial impingement syndrome with glenohumeral internal rotation deficit . Stretching groups will receive either isolytic or static stretching in modified cross body stretching position and standard physiotherapy program. There is a control group. Control group will receive only standard physiotherapy program. Standard physiotherapy program includes TENS, hotpack, posture and strengthening training program. Treatment program will last four times a week (4-4-4-3) for four weeks, 15 sessions in total.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of subacromial impingement syndrome
* Glenohumeral internal rotation range of motion of the affected shoulder should be less than other shoulder and bilateral shoulder internal rotation range of motion difference should be ≥15 º
* Pain with resisted arm elevation or external rotation as well as a minimum of 3 of 5 positive subacromial impingement syndrome tests, painful arc, pain or weakness with resisted external rotation, Neer, Hawkins and Jobe tests.
* Ability to complete the entire study procedure

Exclusion Criteria:

* A 50% limitation of passive shoulder range of motion in >2 planes of motion
* Pain >7/10
* A history of fracture to the shoulder girdle
* Systemic musculoskeletal disease
* History of shoulder and cervical surgery
* Glenohumeral instability (positive apprehension, relocation, or positive sulcus test) or positive findings for a full-thickness rotator cuff tear (positive lag sign, positive drop arm test, or marked weakness with shoulder external rotation)
* Neck and shoulder pain with active/passive cervical spine movement
* A diagnosis of chest deformity or scoliosis
* Regularly performing posterior shoulder stretching exercises

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
Shoulder internal rotation range of motion | Baseline and 4 weeks
  Change of shoulder internal rotation range of motion (with bubble inclinometer)

SECONDARY OUTCOMES:
Glenohumeral internal rotation deficit | Baseline and 4 weeks
  Change of difference in shoulder internal rotation range of motion between the affected and non-affected shoulder (with bubble inclinometer)
Posterior shoulder tightness | Baseline and 4 weeks
  Change of posterior shoulder tightness (with bubble inclinometer)
Shoulder external rotation range of motion | Baseline and 4 weeks
  Change of shoulder external rotation range of motion (with bubble inclinometer)
Shoulder total rotational range of motion | Baseline and 4 weeks
  Change of shoulder total rotational range of motion (Sum of the internal and external rotation motion)
Resting and activitiy pain in shoulder | Baseline and 4 weeks
  Change of visual analog scale score in activity and rest pain
Subacromial space | Baseline and 4 weeks
  Change of subacromial space at arm resting at the side (0°), and at 60° of scapular plane elevation (with Ultrasound)
Supraspinatus tendon thickness | Baseline and 4 weeks
  Change of supraspinatus tendon thickness (with Ultrasound)
Concentric strength | Baseline and 4 weeks
  Change of rotattor cuff muscles concentric strength (in kg, with hand held dynamometer)
Eccentric strength | Baseline and 4 weeks
  Change of shoulder abduction eccentric strength (in kg, with hand held dynamometer)
Shoulder Function | Baseline and 4 weeks
  Change of Modified Constant-Murley Score
Upper extremity function | Baseline and 4 weeks
  Change of disabilities of the arm, shoulder, and hand (Quick-DASH) score

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Sevi YESILYAPRAK, PhD, Study Director — Dokuz Eylul University; Mehmet ERDURAN, MD, Study Director — Dokuz Eylul University; Cem OZCAN, MD, Study Director — Izmır Katip Celebi University Atatürk Training and Research Hospital
Locations (1):
- Dokuz Eylül University, Izmir, Balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No